CLINICAL TRIAL: NCT00677976
Title: Use of Functional Magnetic Resonance Imaging (fMRI) to Study Brain Activation Following Rectal Stimulation in Children With Irritable Bowel Syndrome
Brief Title: Use of Functional Magnetic Resonance Imaging (fMRI) to Study Brain Activation in Children With Irritable Bowel Syndrome
Acronym: fMRI
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Manu Sood, Chief, Associate Professor, Medical College of Wisconsin
Other Study IDs: CHW 06/163
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: fMRI; IBS; Brain Activation
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBS: Children between the ages of 10 and 18 who meet Rome III criteria for IBS as determined by a pediatric gastroenterologist.
- Control: Healthy children between the ages of 10 and 18.

SUMMARY:
The purpose of the study is to map regions of brain activation following rectal stimulation in children with irritable bowel syndrome (IBS) and healthy controls.

DETAILED DESCRIPTION:
Our first aim is to compare the brain areas activated rectal stimulation in boys and girls with IBS and healthy children. Our second aim is to compare the anatomic regions of the brain activated during rectal stimulation in pre and post-pubertal male and female subjects between 10-18 yrs of age.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 years to 18 years who provide written assent and whose parents provide written permission for participation
* English-speaking
* Subjects in the IBS group will meet Rome III criteria for IBS as determined by a pediatric gastroenterologist.

Exclusion Criteria:

* Other pain-related diseases, functional gastrointestinal disorders, or somatization disorder
* Mental retardation or pervasive developmental disorder or epilepsy
* Psychosis
* Genetic or chromosomal disorders
* Currently receiving psychoactive drug treatment
* Patients with pacemakers, metal clips used in previous surgery or other device which are not compatible with MRI scanning
* Inability to lie still in the scanner
* Claustrophobia (Inability to lie still in the scanner)
* Pregnancy
* Subjects who admit to substance abuse during screening
* Orthodontic braces

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children will be selected from the Gastroenterology Clinic at Children's Hospital of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
We intend to measure the degree of brain activation following rectal stimulation | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Manu Sood, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Drossman DA, Li Z, Andruzzi E, Temple RD, Talley NJ, Thompson WG, Whitehead WE, Janssens J, Funch-Jensen P, Corazziari E, et al. U.S. householder survey of functional gastrointestinal disorders. Prevalence, sociodemography, and health impact. Dig Dis Sci. 1993 Sep;38(9):1569-80. doi: 10.1007/BF01303162. PMID 8359066
- [Background] Talley NJ, Zinsmeister AR, Van Dyke C, Melton LJ 3rd. Epidemiology of colonic symptoms and the irritable bowel syndrome. Gastroenterology. 1991 Oct;101(4):927-34. doi: 10.1016/0016-5085(91)90717-y. PMID 1889716
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Hyams JS, Burke G, Davis PM, Rzepski B, Andrulonis PA. Abdominal pain and irritable bowel syndrome in adolescents: a community-based study. J Pediatr. 1996 Aug;129(2):220-6. doi: 10.1016/s0022-3476(96)70246-9. PMID 8765619
- [Background] Hyams JS, Treem WR, Justinich CJ, Davis P, Shoup M, Burke G. Characterization of symptoms in children with recurrent abdominal pain: resemblance to irritable bowel syndrome. J Pediatr Gastroenterol Nutr. 1995 Feb;20(2):209-14. doi: 10.1097/00005176-199502000-00012. PMID 7714688
- [Background] Walker LS, Lipani TA, Greene JW, Caines K, Stutts J, Polk DB, Caplan A, Rasquin-Weber A. Recurrent abdominal pain: symptom subtypes based on the Rome II Criteria for pediatric functional gastrointestinal disorders. J Pediatr Gastroenterol Nutr. 2004 Feb;38(2):187-91. doi: 10.1097/00005176-200402000-00016. PMID 14734882
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Van Ginkel R, Voskuijl WP, Benninga MA, Taminiau JA, Boeckxstaens GE. Alterations in rectal sensitivity and motility in childhood irritable bowel syndrome. Gastroenterology. 2001 Jan;120(1):31-8. doi: 10.1053/gast.2001.20898. PMID 11208711
- [Background] Di Lorenzo C, Youssef NN, Sigurdsson L, Scharff L, Griffiths J, Wald A. Visceral hyperalgesia in children with functional abdominal pain. J Pediatr. 2001 Dec;139(6):838-43. doi: 10.1067/mpd.2001.118883. PMID 11743510
- [Background] Hobson AR, Aziz Q. Brain imaging and functional gastrointestinal disorders: has it helped our understanding? Gut. 2004 Aug;53(8):1198-206. doi: 10.1136/gut.2003.035642. No abstract available. PMID 15247191
- [Background] Aziz Q, Andersson JL, Valind S, Sundin A, Hamdy S, Jones AK, Foster ER, Langstrom B, Thompson DG. Identification of human brain loci processing esophageal sensation using positron emission tomography. Gastroenterology. 1997 Jul;113(1):50-9. doi: 10.1016/s0016-5085(97)70079-9. PMID 9207261
- [Background] Schnitzler A, Ploner M. Neurophysiology and functional neuroanatomy of pain perception. J Clin Neurophysiol. 2000 Nov;17(6):592-603. doi: 10.1097/00004691-200011000-00005. PMID 11151977
- [Background] Willis WD, Westlund KN. Neuroanatomy of the pain system and of the pathways that modulate pain. J Clin Neurophysiol. 1997 Jan;14(1):2-31. doi: 10.1097/00004691-199701000-00002. PMID 9013357
- [Background] Wilder-Smith CH, Schindler D, Lovblad K, Redmond SM, Nirkko A. Brain functional magnetic resonance imaging of rectal pain and activation of endogenous inhibitory mechanisms in irritable bowel syndrome patient subgroups and healthy controls. Gut. 2004 Nov;53(11):1595-601. doi: 10.1136/gut.2003.028514. PMID 15479679
- [Background] Sidhu H, Kern M, Shaker R. Absence of increasing cortical fMRI activity volume in response to increasing visceral stimulation in IBS patients. Am J Physiol Gastrointest Liver Physiol. 2004 Aug;287(2):G425-35. doi: 10.1152/ajpgi.00490.2003. PMID 15246969
- [Background] Lawal A, Kern M, Sanjeevi A, Hofmann C, Shaker R. Cingulate cortex: a closer look at its gut-related functional topography. Am J Physiol Gastrointest Liver Physiol. 2005 Oct;289(4):G722-30. doi: 10.1152/ajpgi.00016.2005. PMID 16160081
- [Background] Drossman DA, Ringel Y, Vogt BA, Leserman J, Lin W, Smith JK, Whitehead W. Alterations of brain activity associated with resolution of emotional distress and pain in a case of severe irritable bowel syndrome. Gastroenterology. 2003 Mar;124(3):754-61. doi: 10.1053/gast.2003.50103. PMID 12612913
- [Background] Derbyshire SW. A systematic review of neuroimaging data during visceral stimulation. Am J Gastroenterol. 2003 Jan;98(1):12-20. doi: 10.1111/j.1572-0241.2003.07168.x. PMID 12526930
- [Background] Lawal A, Kern M, Sidhu H, Hofmann C, Shaker R. Novel evidence for hypersensitivity of visceral sensory neural circuitry in irritable bowel syndrome patients. Gastroenterology. 2006 Jan;130(1):26-33. doi: 10.1053/j.gastro.2005.10.020. PMID 16401465
- [Background] Verne GN, Himes NC, Robinson ME, Gopinath KS, Briggs RW, Crosson B, Price DD. Central representation of visceral and cutaneous hypersensitivity in the irritable bowel syndrome. Pain. 2003 May;103(1-2):99-110. doi: 10.1016/s0304-3959(02)00416-5. PMID 12749964
- [Background] Whitehead WE, Palsson OS. Is rectal pain sensitivity a biological marker for irritable bowel syndrome: psychological influences on pain perception. Gastroenterology. 1998 Nov;115(5):1263-71. doi: 10.1016/s0016-5085(98)70099-x. PMID 9797383
- [Background] Gregory LJ, Yaguez L, Williams SC, Altmann C, Coen SJ, Ng V, Brammer MJ, Thompson DG, Aziz Q. Cognitive modulation of the cerebral processing of human oesophageal sensation using functional magnetic resonance imaging. Gut. 2003 Dec;52(12):1671-7. doi: 10.1136/gut.52.12.1671. PMID 14633941
- [Background] Devinsky O, Morrell MJ, Vogt BA. Contributions of anterior cingulate cortex to behaviour. Brain. 1995 Feb;118 ( Pt 1):279-306. doi: 10.1093/brain/118.1.279. PMID 7895011
- [Background] Paus T. Primate anterior cingulate cortex: where motor control, drive and cognition interface. Nat Rev Neurosci. 2001 Jun;2(6):417-24. doi: 10.1038/35077500. PMID 11389475
- [Background] Rainville P, Duncan GH, Price DD, Carrier B, Bushnell MC. Pain affect encoded in human anterior cingulate but not somatosensory cortex. Science. 1997 Aug 15;277(5328):968-71. doi: 10.1126/science.277.5328.968. PMID 9252330
- [Background] Andresen V, Bach DR, Poellinger A, Tsrouya C, Stroh A, Foerschler A, Georgiewa P, Zimmer C, Monnikes H. Brain activation responses to subliminal or supraliminal rectal stimuli and to auditory stimuli in irritable bowel syndrome. Neurogastroenterol Motil. 2005 Dec;17(6):827-37. doi: 10.1111/j.1365-2982.2005.00720.x. PMID 16336498
- [Background] Lorenz J, Minoshima S, Casey KL. Keeping pain out of mind: the role of the dorsolateral prefrontal cortex in pain modulation. Brain. 2003 May;126(Pt 5):1079-91. doi: 10.1093/brain/awg102. PMID 12690048
- [Background] Vogt BA, Wiley RG, Jensen EL. Localization of Mu and delta opioid receptors to anterior cingulate afferents and projection neurons and input/output model of Mu regulation. Exp Neurol. 1995 Oct;135(2):83-92. doi: 10.1006/exnr.1995.1069. PMID 7589327
- [Background] Kern MK, Jaradeh S, Arndorfer RC, Jesmanowicz A, Hyde J, Shaker R. Gender differences in cortical representation of rectal distension in healthy humans. Am J Physiol Gastrointest Liver Physiol. 2001 Dec;281(6):G1512-23. doi: 10.1152/ajpgi.2001.281.6.G1512. PMID 11705757
- [Background] Berman S, Munakata J, Naliboff BD, Chang L, Mandelkern M, Silverman D, Kovalik E, Mayer EA. Gender differences in regional brain response to visceral pressure in IBS patients. Eur J Pain. 2000;4(2):157-72. doi: 10.1053/eujp.2000.0167. PMID 10957697
- [Background] Naliboff BD, Berman S, Chang L, Derbyshire SW, Suyenobu B, Vogt BA, Mandelkern M, Mayer EA. Sex-related differences in IBS patients: central processing of visceral stimuli. Gastroenterology. 2003 Jun;124(7):1738-47. doi: 10.1016/s0016-5085(03)00400-1. PMID 12806606
- [Background] Houghton LA, Lea R, Jackson N, Whorwell PJ. The menstrual cycle affects rectal sensitivity in patients with irritable bowel syndrome but not healthy volunteers. Gut. 2002 Apr;50(4):471-4. doi: 10.1136/gut.50.4.471. PMID 11889064
- [Background] Berkley KJ. Sex differences in pain. Behav Brain Sci. 1997 Sep;20(3):371-80; discussion 435-513. doi: 10.1017/s0140525x97221485. PMID 10097000
- [Background] Houghton LA, Jackson NA, Whorwell PJ, Morris J. Do male sex hormones protect from irritable bowel syndrome? Am J Gastroenterol. 2000 Sep;95(9):2296-300. doi: 10.1111/j.1572-0241.2000.02314.x. PMID 11007231
- [Background] Chang L, Heitkemper MM. Gender differences in irritable bowel syndrome. Gastroenterology. 2002 Nov;123(5):1686-701. doi: 10.1053/gast.2002.36603. PMID 12404243
- [Background] Petersen S, Bergstrom E, Brulin C. High prevalence of tiredness and pain in young schoolchildren. Scand J Public Health. 2003;31(5):367-74. doi: 10.1080/14034940210165064. PMID 14555373
- [Background] Groholt EK, Stigum H, Nordhagen R, Kohler L. Recurrent pain in children, socio-economic factors and accumulation in families. Eur J Epidemiol. 2003;18(10):965-75. doi: 10.1023/a:1025889912964. PMID 14598927
- [Background] Perquin CW, Hunfeld JA, Hazebroek-Kampschreur AA, van Suijlekom-Smit LW, Passchier J, Koes BW, van der Wouden JC. The natural course of chronic benign pain in childhood and adolescence: a two-year population-based follow-up study. Eur J Pain. 2003;7(6):551-9. doi: 10.1016/S1090-3801(03)00060-0. PMID 14575668
- [Background] Chitkara DK, Rawat DJ, Talley NJ. The epidemiology of childhood recurrent abdominal pain in Western countries: a systematic review. Am J Gastroenterol. 2005 Aug;100(8):1868-75. doi: 10.1111/j.1572-0241.2005.41893.x. PMID 16086724
- [Background] Hunfeld JA, Perquin CW, Hazebroek-Kampschreur AA, Passchier J, van Suijlekom-Smit LW, van der Wouden JC. Physically unexplained chronic pain and its impact on children and their families: the mother's perception. Psychol Psychother. 2002 Sep;75(Pt 3):251-60. doi: 10.1348/147608302320365172. PMID 12396752
- [Background] Caviness VS Jr, Kennedy DN, Richelme C, Rademacher J, Filipek PA. The human brain age 7-11 years: a volumetric analysis based on magnetic resonance images. Cereb Cortex. 1996 Sep-Oct;6(5):726-36. doi: 10.1093/cercor/6.5.726. PMID 8921207
- [Background] Reiss AL, Abrams MT, Singer HS, Ross JL, Denckla MB. Brain development, gender and IQ in children. A volumetric imaging study. Brain. 1996 Oct;119 ( Pt 5):1763-74. doi: 10.1093/brain/119.5.1763. PMID 8931596
- [Background] Giedd JN, Snell JW, Lange N, Rajapakse JC, Casey BJ, Kozuch PL, Vaituzis AC, Vauss YC, Hamburger SD, Kaysen D, Rapoport JL. Quantitative magnetic resonance imaging of human brain development: ages 4-18. Cereb Cortex. 1996 Jul-Aug;6(4):551-60. doi: 10.1093/cercor/6.4.551. PMID 8670681
- [Background] Burgund ED, Kang HC, Kelly JE, Buckner RL, Snyder AZ, Petersen SE, Schlaggar BL. The feasibility of a common stereotactic space for children and adults in fMRI studies of development. Neuroimage. 2002 Sep;17(1):184-200. doi: 10.1006/nimg.2002.1174. PMID 12482076
- [Background] Kang HC, Burgund ED, Lugar HM, Petersen SE, Schlaggar BL. Comparison of functional activation foci in children and adults using a common stereotactic space. Neuroimage. 2003 May;19(1):16-28. doi: 10.1016/s1053-8119(03)00038-7. PMID 12781724
- [Background] Duke PM, Litt IF, Gross RT. Adolescents' self-assessment of sexual maturation. Pediatrics. 1980 Dec;66(6):918-20. PMID 7454482
- [Derived] Liu X, Li SJ, Shaker R, Silverman A, Kern M, Ward DB, Li W, Xu Z, Chelimsky G, Sood MR. Reduced Functional Connectivity Between the Hypothalamus and High-order Cortical Regions in Adolescent Patients With Irritable Bowel Syndrome. J Pediatr Gastroenterol Nutr. 2017 Nov;65(5):516-519. doi: 10.1097/MPG.0000000000001611. PMID 29064927